CLINICAL TRIAL: NCT04773002
Title: A Comparison of Volatile Anesthesia and Total Intravenous Anesthesia (TIVA) on Ecchymosis, Edema, and Intraoperative Bleeding in Rhinoplasty
Brief Title: A Comparison of Volatile Anesthesia and Total Intravenous Anesthesia (TIVA)
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hakan Tapar, Associate professor, Tokat Gaziosmanpasa University
Other Study IDs: 21-KAEK-006
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Rhinoplasty; Ecchymosis; Edema; Hemorrhage
MeSH Terms: conditions — Ecchymosis; Edema; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: Total intravenous anesthesia (TIVA)
  Interventions: Other: Different anesthesia methods
- Group S: Volatile anestesia
  Interventions: Other: Different anesthesia methods

INTERVENTIONS:
Other: Different anesthesia methods — Total intravenous anesthesia (TIVA)and volatile anesthesia

SUMMARY:
In this study, investigators wanted to investigate the effect of volatile anesthesia and total intravenous anesthesia (TIVA) on ecchymosis, edema, and intraoperative bleeding in rhinoplasty.

DETAILED DESCRIPTION:
Routine monitorization (blood pressure, pulse, oxygen saturation with pulse oximetry and electrocardiogram) will be applied to all patients taken into the operation room.

In Group P (TIVA), induction of anesthesia will be achieved with 2 mg/kg propofol, 0.6 mg/kg rocuronium, and 1 μ / kg fentanyl. Propofol and remifentanil will be used in the continuation of anesthesia.

In Group S (Volatile), anesthesia will be induced with 2 mg / kg propofol, 0.6 mg / kg rocuronium and 1 μ / kg fentanyl. 50% nitrous oxide + 50% oxygen and 2% sevoflurane will be used in the continuation of anesthesia.

All patients will receive 2 ml/kg/hour Ringer's lactate solution during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years
* Planned to rhinoplasty
* An American Society of Anesthesiologists score of 1 or 2

Exclusion Criteria:

* Steroid use
* Patients with coagulation disorders, •Rejected to participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rhinoplasty patients
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-08-21 (Actual)

PRIMARY OUTCOMES:
Edema and ecchymosis in rhinoplasty according to the type of anesthesia. | one time in six months
  It is evaluation developing edema and ecchymosis according to total intravenous anesthesia and volatile anesthesia in rhinoplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Katar, Study Chair — Gaziosmanpasa university
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)